CLINICAL TRIAL: NCT01055197
Title: Randomized Phase II Study Comparing Prophylactic Cranial Irradiation Alone to Prophylactic Cranial Irradiation and Consolidative Extra-Cranial Irradiation for Extensive Disease Small Cell Lung Cancer (ED-SCLC)
Brief Title: Radiation Therapy in Treating Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0937; CDR0000663959; NCI-2011-02008 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI (Experimental): Prophylactic Cranial Irradiation (PCI)
  Interventions: Radiation: Prophylactic Cranial Irradiation
- PCI + Consolidation RT (Experimental): Prophylactic Cranial Irradiation (PCI) plus consolidative radiation therapy (RT) to locoregional and residual metastatic disease
  Interventions: Radiation: Prophylactic Cranial Irradiation; Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation — Prophylactic Cranial Irradiation (PCI) to the brain in ten once-daily fractions of 2.5 Gy, five days per week, for a total of 25 Gy.
  Other Names: PCI
Radiation: Radiation Therapy — Radiation Therapy (RT) to locoregional and residual metastatic disease in 15 once daily fractions of 3.0 Gy, 5 days per week, for a total of 45 Gy
  Other Names: RT
  Arms: PCI + Consolidation RT

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. This may be an effective treatment for extensive stage small cell lung cancer.

PURPOSE: This randomized phase II trial is comparing how well radiation therapy to the brain works when given with or without radiation therapy to other areas of the body in treating patients with extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the 1-year overall median survival rate in patients with extensive stage small cell lung cancer treated with prophylactic cranial irradiation with vs without consolidative extracranial radiotherapy following platinum-based chemotherapy.

Secondary

* To compare treatment-related adverse events in these patients.
* To evaluate patterns of failure in these patients.
* To compare the time to first failure in these patients.
* To evaluate the percentage of the planned radiotherapy dose given to each site.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior treatment (complete response vs partial response) and number of metastatic lesions (1 vs 2-3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo prophylactic cranial irradiation 5 days per week for 2 weeks.
* Arm II: Patients undergo prophylactic cranial irradiation as in arm I. Patients also undergo consolidative extracranial radiotherapy to locoregional and residual metastatic disease 5 days per week for 2-3 weeks.

After completion of study treatment, patients are followed up at 2 weeks; at 1, 2, 6, 9, and 12 months; every 6 months for 2 years; and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed extensive stage small cell lung cancer (SCLC) diagnosed within the past 6 months*

  * Has 1-4 extracranial metastatic lesions NOTE: *Diagnosis made before treatment with chemotherapy
* Has completed 4-6 courses of platinum-based chemotherapy within the past 8 weeks AND meets the following criteria:

  * Radiographic partial or complete response to chemotherapy in ≥ 1 site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria (if radiotherapy has been delivered to primary disease with chemotherapy, there must be complete or partial response in ≥ 1 of the sites that has not been treated with radiotherapy)
  * No progression in any site
* No limited stage SCLC, even if disease progressed
* No brain or central nervous system (CNS) metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Platelets ≥ 75,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (the use of transfusion or other intervention is allowed)
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN) (for patients who will receive radiotherapy to the liver)
* Serum bilirubin < 1.5 times ULN (for patients who will receive radiotherapy to the liver)
* Serum creatinine < 1.5 times ULN (for patients who will receive radiotherapy to the kidneys)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe, active co-morbidity, defined as any of the following:

  * Acute bacterial or fungal infection requiring IV antibiotics at the time of study registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of study registration

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior chemotherapy (i.e., toxicities ≤ grade 1 [except for neuropathy and alopecia])
* Thoracic radiotherapy administered concurrently with or before chemotherapy for the current diagnosis allowed (these patients will not receive mediastinal radiotherapy per protocol)
* No prior radiotherapy to the region of this cancer that would result in overlap of radiotherapy fields
* No concurrent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Gore, MD, Principal Investigator — Medical College of Wisconsin; Alexander Sun, MD, Principal Investigator — Princess Margaret Cancer Center
Locations (115):
- United States (108):
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Saint Agnes Cancer Center at Saint Agnes Medical Center, Fresno, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology, PA at Texas Cancer Center - Arlington South, Arlington, Texas
  - Texas Oncology, PA at Texas Cancer Center - Denton South, Denton, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Hospital - Memorial City, Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - Cancer Care Centers of South Texas - Northeast, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology, PA - Wichita Falls, Wichita Falls, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
- Canada (5):
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- Israel (2):
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic Cranial Irradiation: Prophylactic Cranial Irradiation (PCI)
- Prophylactic Cranial Irradiation + Consolidation Radiotherapy: Prophylactic Cranial Irradiation (PCI) plus consolidative radiation therapy (RT) to locoregional and residual metastatic disease
Period: Overall Study
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Started | 51 | 46
Completed | 42 (Subjects with data available for the primary analysis are considered to have completed the study.) | 44 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 9 | 2
Not completed — Protocol Violation | 7 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 81] | 66 [35 to 86] | 63 [35 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (12-month Rate Reported)
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur when all patients had been potentially followed for at least 12 months. The 12-month rate is reported.
Time Frame: From randomization to last follow-up. Analysis occurred after all patients had been potentially followed for at least 12 months. Maximum follow-up at time of analysis was 46.0 months.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Number analyzed (Participants) | 42 | 44
percentage of participants | 60.1 [41.2 to 74.7] | 50.8 [34.0 to 65.3]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation vs Prophylactic Cranial Irradiation + Consolidation Radiotherapy; The null hypothesis (H0) was that PCI + RT is not effective versus the alternative hypothesis (H1) that PCI + RT is effective. Assumptions were that PCI alone would have hazard rate λc of 1.204 and PCI + RT a hazard rate λc of 0.799 (hazard ratio λt/λc = 0.663). At each planned analysis, the p-value from the log-rank test statistic assessing overall survival was compared to the nominal significance level. The final targeted accrual was 154; Test type: Superiority or Other; p = 0.2103, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.82 to 2.53]

2. Secondary Outcome: Percentage of Patients Experiencing a Grade 3 or Higher Adverse Event
Description: Adverse events (AE) are graded using CTCAE v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: as for outcome 1
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Number analyzed (Participants) | 42 | 44
percentage of participants | 24 [12 to 39] | 36 [22 to 52]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation vs Prophylactic Cranial Irradiation + Consolidation Radiotherapy; Test type: Superiority; p = 0.24, Fisher Exact; 2-sided significance level of 0.05

3. Secondary Outcome: Patterns of Failure - Number of Patients With Failure by Site
Description: Failure was defined as progressive disease in areas treated with radiation development of measurable disease at sites that had achieved a complete response either with chemotherapy prior to study entry or following radiation, or development of new disease characteristic of small-cell lung cancer dissemination as determined by imaging [per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1] and physical examination. A patient could be counted in more than one category.
Time Frame: as for outcome 1
Population: All eligible patients who had a failure
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Number analyzed (Participants) | 32 | 31
Participants
  1st failure site = diagnosis site | 25 | 13
  1st failure site = locoregional disease | 20 | 8
  1st failure site = brain | 0 | 6
  Failure at any time at new site | 10 | 19

4. Secondary Outcome: First Failure (12-month Rate Reported)
Description: Failure was defined as progressive disease in areas treated with radiation development of measurable disease at sites that had achieved a complete response either with chemotherapy prior to study entry or following radiation, or development of new disease characteristic of small-cell lung cancer dissemination as determined by imaging [per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1] and physical examination. Time to first failure is defined as time from randomization to the date of first failure, last known follow-up (censored), or death (competing risk). First failure rates are estimated using the cumulative incidence method.
Time Frame: as for outcome 1
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Number analyzed (Participants) | 42 | 44
percentage of participants | 79.6 [60.6 to 90.2] | 75.0 [57.9 to 86.0]
Statistical Analysis 1: Comparison: Prophylactic Cranial Irradiation vs Prophylactic Cranial Irradiation + Consolidation Radiotherapy; Test type: Superiority; p = 0.0102, Log Rank; 2-sided significance level of 0.05

5. Secondary Outcome: Percentage of Planned Radiotherapy Dose (All Sites) That Was Delivered
Description: Total dose to the brain was to be 25 Gy for all patients. For patients on PCI+consolidative RT, patients were to get 45 Gy at 3 Gy per fraction to the locoregional area as well as to residual metastatic disease. Alternatively, these regions could have received 30-40 Gy in 10 fractions. The total planned dose was determined, and a percentage was calculated based for each patient as total delivered dose / total planned dose.
Time Frame: From start to end of radiation therapy; up to 32 days for Prophylactic Cranial Irradiation arm, up to 68 days for Prophylactic Cranial Irradiation + Consolidation Radiotherapy arm.
Population: All eligible patients who started study treatment
Measure: Median (Full Range); unit: percentage of planned dose delivered
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Number analyzed (Participants) | 42 | 44
percentage of planned dose delivered | 100 [70 to 100] | 100 [62 to 115]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Prophylactic Cranial Irradiation | Prophylactic Cranial Irradiation + Consolidation Radiotherapy
Serious Adverse Events (participants affected / at risk) | 1/42 | 6/44
Other Adverse Events (participants affected / at risk) | 37/42 | 36/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylactic Cranial Irradiation (N=42) | Prophylactic Cranial Irradiation + Consolidation Radiotherapy (N=44)
Sinus tachycardia (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylactic Cranial Irradiation (N=42) | Prophylactic Cranial Irradiation + Consolidation Radiotherapy (N=44)
Anemia (Blood and lymphatic system disorders) | 7 | 9
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 3 | 1
Blurred vision (Eye disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 6 | 10
Dyspepsia (Gastrointestinal disorders) | 4 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 11
Nausea (Gastrointestinal disorders) | 16 | 14
Vomiting (Gastrointestinal disorders) | 8 | 3
Fatigue (General disorders) | 27 | 26
Pain (General disorders) | 5 | 6
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 | 6
Platelet count decreased (Investigations) | 3 | 5
Weight loss (Investigations) | 8 | 10
Anorexia (Metabolism and nutrition disorders) | 6 | 19
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 5
Dysgeusia (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 17 | 6
Memory impairment (Nervous system disorders) | 5 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 5 | 4
Depression (Psychiatric disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
At the first interim analysis of overall survival the data monitoring committee determined that due to the lack of evidence of potential efficacy and a higher than acceptable toxicity profile for the PCI+RT arm, study accrual would close early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.